CLINICAL TRIAL: NCT01830426
Title: Phase 2 Study of Circulating Tumor Cell in Non-Small Cell Lung Carcinoma
Brief Title: Circulating Tumor Cells in Non-Small Cell Lung Carcinoma
Acronym: LDx
Status: Completed | Type: Observational
Sponsor: Epic Sciences (Industry)
Collaborators: Yale University (Other); Billings Clinic (Other); University of California, San Diego (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: HHSN261201200049C; HHSN26120100049C (Other Grant/Funding Number: National Cancer Institute)
Record Dates: First submitted 2013-03-25; First posted 2013-04-12 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Primary Lung Cancer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cell solution plated onto slides and frozen for storage
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to establish the circulating tumor cell (CTC) assay as a surrogate for tissue diagnosis of suspected primary lung cancer. This is done through evaluating clinical and molecular markers to stratify the outcome/survival in patients with thoracic malignancies treated at Yale University/Yale-New Haven Hospital, University of California San Diego/Moores Cancer Center, Billings Clinic Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

* Suspected lung cancer
* Planned to undergo tissue biopsy. Tissue biopsy does not need to be limited to an intrathoracic structures. Biopsies of the supraclavicular lymph nodes are allowed
* Age >18

Exclusion Criteria:

* Patients with history of a separate (not a primary lung cancer) malignancy within past two years.
* Recent history (past two weeks) of trauma (INCLUDING diagnostic surgery, biopsy, etc)
* Prior lung cancer treatment chemotherapy, radiation, surgery, etc. in past two years.
* Inability to provide informed consent.
* Hgb less than 8.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A primary lung cancer bearing population will be studied. Eligible patients will include those presenting to the specified clinical centers with a tissue confirmed primary lung cancer or radiographic abnormality deemed highly suspicious for primary lung cancer by collaborating clinical team, in whom definitive tissue diagnosis is planned. All stages of primary lung cancer will considered.
Sampling Method: Non-Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2012-11; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
CTC Enumeration | 3 months from baseline, an average of 2 weeks post patient tissue biopsy
  After informed consent of the patients, a single tube of blood will be drawn and processed according to the standard protocol. These blood draws will occur upon patient screening or rather the baseline of their treatment, a 6-12 week follow-up, as well as a 12 month follow-up.Furthermore, a biopsy will be taken between baseline and 6-12 week follow-up which will be used upon results of CTC enumeration to illustrate concordance. Epic Sciences staff is fully blinded to the clinical data of the patients until final analysis. Patients will be considered CTC positive at a count of greater than 2 CTCs per ml of blood.

SECONDARY OUTCOMES:
Lung Cancer Subtyping | 3 months from baseline, an average of 2 weeks post patient tissue biopsy
  Based on the blood draws from the primary outcome, Epic will utilize the identified CTCs as biopsy material for lung cancer subtyping that distinguishes between adenocarcinoma (ACA), squamous cell carcinoma (SCC) from other types of primary lung cancer. Lung cancer histology will be evaluated for each patient sample: Two slides will be run with the ACA-CTC assay (TTF1 or Napsin A) and two slides will be run with the SCC-CTC (p63) assay. For the purpose of assay development and validation, we have all already procured a validated set of patient samples with known histology.
Nodal Staging | 3 months from baseline, an average of 2 weeks post patient tissue biopsy
  For patients ultimately diagnosed with lung cancer and deemed to be surgical candidates, surgical intervention will be performed. In accordance to a standard practice mediastinal lymph node dissection will accompany the surgery. Nodal staging for each patient in the trial with diagnosed lung cancer will be evaluated clinically and pathologically. Clinical staging will be determined by the treating clinician prior to information being available from surgery and recorded in the case report form. The diagnostic accuracy of the clinical stage will be determined by comparison with the pathological stage which will be abstracted from the pathology report for surgically staged patients. We will determine the sensitivity and specificity of the CTC count as a test that identifies patients who will ultimately be "upstaged" from N0 to N1 or from N1 to N2-3 at the time of surgical staging when comparing the clinical and pathological stage.
Establish the Prognostic Value by measuring CTC count over time. | Baseline, 3 months, 24 months and 66 months
  This measure will work to establish the prognostic value of the initial test by drawing the correlation with outcome data. For the 260 patients recruited to this clinical trial, stage specific Kaplan-Meier overall and disease free survival curves for the population will be generated after 2 years of follow-up. For each stage, the results of the CTCs will then be used to separate the population for each stage into a low CTC and high CTC group to determine if the disease free survival curves for each stage separate on the basis of the assay and are statistically significant using a retrospective analysis of the prospectively collected data, this will determine if knowledge of the CTC assay provides useful information about disease free survival beyond that which is obtained by clinical staging alone.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Dittamore, MBA, Principal Investigator — Epic Sciences
Locations (3):
- United States (3):
  - Moores Cancer Center, La Jolla, California
  - Yale University, New Haven, Connecticut
  - Billings Clinic Cancer Center, Billings, Montana